CLINICAL TRIAL: NCT00006057
Title: Diagnostic and Screening Study of Genetic Disorders
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: 199/15151; MTS-GCO-88-459
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Tay-Sachs Disease; Porphyria, Erythropoietic; Leukodystrophy, Globoid Cell; Metabolism, Inborn Errors
MeSH Terms: conditions — Tay-Sachs Disease; Porphyria, Erythropoietic; Leukodystrophy, Globoid Cell; Metabolism, Inborn Errors

SUMMARY:
OBJECTIVES: I. Determine the phenotypic heterogeneity of patients with genetic disorders including their clinical spectrum and natural history.

II. Develop and evaluate novel methods for the treatment of genetic disorders including metabolic manipulation, enzyme manipulation, enzyme replacement, enzyme transplantation, and gene transfer techniques in these patients.

III. Develop and evaluate methods for the prenatal diagnosis of genetic disorders using improved cytogenetic, biochemical, and nucleic acid techniques and amniotic fluid cells or chorionic villi in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are evaluated annually or biannually, depending on disease status and progression. Patients undergo a complete medical history, an extensive family pedigree, and a physical examination. Patients undergo general laboratory, imaging, physiologic, and clinical laboratory studies according to their disease type. Patients undergo specialized laboratory studies including plasma and leukocyte enzyme assays, quantitative urinary mucopolysaccharides and oligosaccharides, urine and plasma glycolipids, plasma and urine amino acids, urine organic acids, lymphoblastoid culture, DNA isolation from peripheral leukocytes, skin biopsy for fibroblast culture (if indicated), and medical photography. Patients also receive consultations with various specialties including ophthalmology, ENT, cardiology, pulmonary, gastroenterology/nutrition, hematology, neurology, orthopedics, rehabilitation medicine/physical therapy, and dermatology.

ELIGIBILITY:
* Suspected diagnosis (homozygous or heterozygous) of a genetic disorder including, but not limited to, one of the following: Tay-Sachs disease (adult form) Congenital erythropoietic porphyria Galactosemia Mitochondrial myopathy Globoid cell leukodystrophy (Krabbe disease) Methylmalonic acidemia Isovaleric acidemia Morquio type A Glycogen storage disease type 1AB Ornithine aminotransferase deficiency Ceroid lipofuscinosis Glutaric aciduria type 1 Citrullinemia Other malformation syndromes, lysosomal storage disorders, or peroxisomal disorders

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Judith P. Willner, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States